CLINICAL TRIAL: NCT04508842
Title: The Phase I Efficacy and Safety Clinical Study of CD19/CD22-Dual-STAR-T Cells in Relapsed and Refractory B-ALL.
Brief Title: CD19/CD22-Dual-STAR-T for Patients With B Cell Acute Leukemia(B-ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment plan
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-011
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-05

CONDITIONS: Refractory and Relapsed B Cell Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD22-Dual-STAR-T (Experimental): CD19/CD22-Dual-STAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of Dual-STAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 500mg/m2 for 3 days and take a rest for 2 days before infusion. Dual-STAR-T cells will be intravenously infused with a escalated dose of 6E5、1E6、2E6、3E6 cells/kg.
  Interventions: Biological: CD19/CD22-Dual-STAR-T

INTERVENTIONS:
Biological: CD19/CD22-Dual-STAR-T — Patients with B cell acute leukemia will be enrolled, and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of CD19/CD22-Dual-STAR-T cells.Dual-STAR-T cells will be intravenously infused with a escalated dose of 6E5、1E6、2E6、3E6 cells/kg.

SUMMARY:
This is a single center, single arm, open-lable phase I study to determine the safety and efficacy of CD19/CD22-Dual-STAR-T cells in patients with refractory and relapsed B cell acute leukemia .

DETAILED DESCRIPTION:
Patients with B cell acute leukemia will be enrolled, and Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of Dual-STAR-T cells.Dual-STAR-T cells will be intravenously infused with a escalated dose of 6E5、1E6、2E6、3E6 cells/kg.The purpose of current study is to evaluate the clinical safety and efficacy of CD19/CD22-Dual-STAR-T cells therapy in patients with refractory and relapsed B-ALL.Safety and efficacy of Dual-STAR-T cells therapy will be monitored. The primary endpoint is the safety of Dual-STAR-T cells including the effect ratio of CRS and ICANS, ORR. The secondary endpoint is the Dual-STAR-T cell proliferation ratio and Dual-STAR gene copied number in peripheral blood（PB）， and progression free survival(PFS ), overall-survival(OS) and duration of overall response(DOR).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 1 to 70 years.
2. Prelapsed and refractorys B-ALL at least with one of the following conditions:

   * Could not achieve CR after 2course of chemotherapy.
   * Could not achieve CR or relapse after first-line or multi-line salvage chemotherapy, or MRD≥0.1%.
   * Relapse within 12 months after first remission or MRD≥0.1%.
   * Relapse after achieved CR in allogeneic hematopoietic stem cell transplantation (HSCT), or MRD≥0.1%.
   * For Ph + patients: Failure to tolerate TKI or TKI treatment failure could be enrolled.
3. CD19 and/or CD22 positive within 3 months.
4. ECOG 0-2.
5. Estimated life expectancy ≥ 3 months.
6. Women of childbearing age must receive a pregnancy test within 7 days prior to initiation of treatment and the results are negative; male and female patients with fertility must use an effective contraceptive to ensure 12 months after discontinuation of treatment during the study period not pregnant inside.
7. Patients who voluntarily sign informed consent and are willing to comply with treatment plans, visit arrangements, laboratory tests and other research procedures.

Exclusion Criteria:

1. Active infections that are difficult to control
2. HBV-DNA HCV-RNA and HIV ,either of which is positive
3. Central nervous system leukemias that is symptomatic or uncontrolled by systemic chemotherapy and intrathecal chemotherapy
4. Patients are receiving anti-GVHD treatment within 4 weeks of before screening.
5. Performed major surgery within 4 weeks before screening.
6. Patients have received chemotherapy within 7 days of screening.
7. Experimental drugs were used within 4 weeks before screening.
8. Received allogeneic cell therapy within 6 weeks prior to cell infusion.
9. Patients have history of epilepsy or central nervous system diseases.
10. Severe thyroid dysfunction
11. Patients with active autoimmune disease.
12. Pregnant or lactating women.
13. The patient does not agree to use effective contraception during treatment and for the following 12 months;
14. The researchers found that it was unsuitable for the recipients to be enrolled.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events. | 12 months
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Objective Remission Rate(ORR) | 12 months
  The percentage of participants who achieved complete remission(CR) and CR in over all participants.
Proliferation ratio of Dual-STAR-T cells | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xian Zhang, PhD, Study Director — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China